CLINICAL TRIAL: NCT05040984
Title: Predictors Affecting Long-term Use of Solifenacin or Mirabegron in Women With Overactive Bladder Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief of Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 110053-E
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Overactive Bladder Syndrome
MeSH Terms: interventions — Solifenacin Succinate; mirabegron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- solifenacin
  Interventions: Drug: Solifenacin Oral Tablet
- mirabegron
  Interventions: Drug: Mirabegron 25mg

INTERVENTIONS:
Drug: Solifenacin Oral Tablet — Solifenacin 1 tablet per day
  Groups: solifenacin
Drug: Mirabegron 25mg — Mirabegron 1 tablet per day
  Groups: mirabegron

SUMMARY:
A retrospective analysis of medical records at Far Eastern Memorial Hospital from January 2008 to May 2020 about female patients with overactive bladder syndrome, who received Solifenacin or Mirabegron as the initial treatment. Factors affecting persistence of OAB medications will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Women with overactive bladder syndrome received solifenacin or mirabegron as the initial treatment

Exclusion Criteria:

* <20 year-old

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women with overactive bladder syndrome, who received Solifenacin or Mirabegron as the initial treatment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictors of persistence of mirabegron versus solifenacin use | 13 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan